CLINICAL TRIAL: NCT00099229
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Tolerability of Licarbazepine 1000-2000mg/Day in the Treatment of Manic Episodes of Bipolar I Disorder Over 3 Weeks
Brief Title: Study of Licarbazepine in the Treatment of Manic Episodes of Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIC477D2301
Record Dates: First submitted 2004-12-10; First posted 2004-12-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; manic episode; treatment; licarbazepine
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

INTERVENTIONS:
Drug: Licarbazepine

SUMMARY:
This purpose of this study is to evaluate the safety and efficacy of Licarbazepine for the treatment of manic episodes of bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder (type I) with manic or mixed episodes (including patients with/without psychotic features or with/without a history of rapid cycling)
* In need of psychiatric treatment
* Cooperation and willingness to complete all aspects of the study

Exclusion Criteria:

* Current diagnosis other than bipolar I disorder
* History of schizophrenia or schizoaffective disorder
* Drug dependence within 1 month prior to study start or testing positive in a urine drug test
* Suicide attempt within 1 month prior to study start or at immediate risk of harm to self or others
* Any form of psychotherapy within 1 month prior to study start

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2004-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Mean reduction in manic episodes and major depressive episodes from baseline to endpoint (Week 3).

SECONDARY OUTCOMES:
Major improvement in anxiety and depression from baseline to endpoint (Week 3)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (15):
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Cerritos, California
  - Investigational Site, San Diego, California
  - Investigational Site, Port Charlotte, Florida
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Newton, Kansas
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Raleigh, North Carolina
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Austin, Texas
  - Investigational Site, Bellaire, Texas
  - Investigational Site, Houston, Texas
  - Investigational Site, Kirkland, Washington
- France (2):
  - Investigational Site, Dijon
  - Investigational Site, Strasbourg
- Russia (2):
  - Investigational Site, Moscow
  - Investigational Site, Saint Petersburg

REFERENCES:
- See also: Click here for further information and to find an investigational site near you — http://www.novartisclinicaltrials.com/etrials/DiseaseID10/Bipolar-Disorder-clinical-trials.go